CLINICAL TRIAL: NCT04293341
Title: A Comparison of the Efficacy of Transdiagnostic Behavior Therapy and Disorder-specific Therapy in Veterans With PTSD, Anxiety, and Depression
Brief Title: Comparing Individual Therapies for Veterans With Depression, PTSD, and Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBB-005-19S
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder; Posttraumatic Stress Disorder; Panic Disorder and Agoraphobia
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Panic Disorder; Agoraphobia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdiagnostic Behavior Therapy (Experimental): TBT was developed to address transdiagnostic avoidance via the use of four different types of exposure techniques (situational/in-vivo, physical/interoceptive, thought/imaginal, and [positive] emotional/behavioral activation). From the transdiagnostic avoidance perspective, the four exposure practices are matched to the type(s) of avoidance experienced by patients based upon their cluster of symptoms/disorders.
  Interventions: Behavioral: Transdiagnostic Behavior Therapy
- Disorder Specific Therapies (Active Comparator): To provide an evidence-based comparison for the TBT condition, DSTs will be used that are matched to the participant's most severe diagnosis, based upon the average of the ADIS interference and distress scores. If the scores are equivalent for two or more diagnoses, participants will be asked to list which diagnosis/symptoms that they find most impairing. DSTs will be included for each of the three targeted diagnoses, including PTSD (CPT for PTSD), PD/AG (CBT for PD/AG), and MDD (CBT for MDD). Each of these DSTs have published manuals for administration and have received extensive support in the literature (Barlow, 2014).
  Interventions: Behavioral: Cognitive Processing Therapy for PTSD; Behavioral: Cognitive Behavioral Therapy for MDD; Behavioral: Cognitive Behavioral Therapy for Panic Disorder

INTERVENTIONS:
Behavioral: Transdiagnostic Behavior Therapy — TBT was developed to address transdiagnostic avoidance via the use of four different types of exposure techniques (situational/in-vivo, physical/interoceptive, thought/imaginal, and [positive] emotional/behavioral activation). From the transdiagnostic avoidance perspective, the four exposure practices are matched to the type(s) of avoidance experienced by patients based upon their cluster of symptoms/disorders.
  Arms: Transdiagnostic Behavior Therapy
Behavioral: Cognitive Processing Therapy for PTSD — CPT is a well established evidence-based psychotherapy for PTSD. CPT focuses on teaching patients to evaluate and change the upsetting thoughts that they have had since their trauma.
  Arms: Disorder Specific Therapies
Behavioral: Cognitive Behavioral Therapy for MDD — CBT for MDD is a well established evidence-based psychotherapy for depression. CBT for MDD focuses teaching patients how to change their behaviors and challenge their negative thoughts to improve their mood.
  Arms: Disorder Specific Therapies
Behavioral: Cognitive Behavioral Therapy for Panic Disorder — CBT for Panic Disorder is a well established evidence-based psychotherapy. CBT for Panic Disorder focuses teaching patients how to change their behaviors through exposure practices and challenge their anxious thoughts to reduce their experience of panic attacks and avoidance.
  Arms: Disorder Specific Therapies

SUMMARY:
Cognitive behavioral therapy (CBT) is a brief, efficient, and effective treatment for individuals with depressive/anxiety disorders. However, CBT is largely underutilized within the Department of Veterans Affairs due to the cost and burden of trainings necessary to deliver all of the related disorder-specific treatments (DSTs). Transdiagnostic Behavior Therapy (TBT), in contrast, is specifically designed to address numerous distinct disorders within a single protocol in Veterans with depressive/anxiety disorders, including posttraumatic stress disorder. The proposed research seeks to evaluate the efficacy of TBT by assessing psychiatric symptomatology and related impairment outcomes in Veterans with depressive/anxiety disorders via a randomized controlled trial of TBT and existing DSTs in Veterans with major depressive disorder, posttraumatic stress disorder, and panic disorder. Assessments will be completed at pre-, mid-, and post-treatment, and at 6-month follow-up. Process variables also will be investigated.

DETAILED DESCRIPTION:
Objective To examine efficacy of Transdiagnostic Behavior Therapy (TBT) on improving psychiatric symptomatology and related impairments in Veterans with major depressive disorder (MDD), posttraumatic stress disorder (PTSD), and panic disorder and agoraphobia (PD/AG) compared to disorder-specific treatments (DSTs) via a non-inferiority design. Patient satisfaction and predictors of feasibility (attendance and discontinuation) also will be assessed.

Recruitment Strategy and Feasibility of Recruitment Veterans will be recruited through the Primary Care Mental Health Integration, General Outpatient Mental Health, and CBT Clinic programs at the Ralph H. Johnson VAMC and all affiliated VA community-based outpatient clinics. IRB-approved study flyers will be distributed through each clinic/setting. Within these programs, all Veterans reporting symptoms of depression and anxiety meet with a mental health staff member to complete a clinical interview and self-report measures. If Veterans endorse symptoms consistent with a depressive/anxiety disorder, interest in participating in research will be assessed and, if agreeable, the Veteran will be referred to project staff. A research assessment will be completed with the project staff to first complete consent documentation and then assess inclusion/exclusion criteria (with a targeted sample of 306 VAMC patients), including a semi-structured clinical interview and self-report questionnaires focused on psychiatric symptomatology and related impairments (described later). Participants who meet inclusion/exclusion criteria will be randomized into a study condition and will be assigned to a project therapist. Because most VA Medical Center (VAMC) patients who meet study criteria likely will present with multiple depressive/anxiety disorders, principal diagnosis, or the most impairing of the diagnosable disorders, will be used to inform randomization. Principal diagnosis will be determined via diagnostic severity scores in the Anxiety Disorders Interview Schedule-5 (ADIS-5). To balance diagnoses across the two conditions, a stratified random assignment based on principal diagnosis will be used (MDD, PTSD, and PD/AG).

Procedures Eligible VAMC patients will be randomized into one of two treatment conditions: TBT or DSTs. Both treatment conditions will include 12 weekly 45- to 60-minute treatment sessions. The general format of sessions will involve: 1) brief check-in; 2) review of materials from previous sessions; 3) review of homework assignments; 4) overview of new materials and in-session exercises; and 5) assignment of homework for next session. Attendance and homework completion will be recorded.

Randomization Procedures Participants will be randomly assigned (1:1) to one of the two study arms (n = 108 per arm) using a permuted block randomization procedure. Randomization will be stratified by diagnostic group (PTSD, PD/AG, MDD) and block size will be varied to minimize the likelihood of unmasking. After determining eligibility and completing consent and baseline assessment materials, enrolled participants will be assigned to their treatment condition by the Research Project Therapist/Coordinator using a computer-generated randomization scheme.

Transdiagnostic Behavior Therapy TBT was developed as a streamlined protocol to address transdiagnostic avoidance via the use of four different types of exposure techniques (situational/in-vivo, physical/interoceptive, thought/imaginal, and positive emotional). From the transdiagnostic avoidance perspective, the four exposure practices are matched to the type(s) of avoidance experienced by patients based upon their cluster of symptoms/disorders. Per protocol, the first six sessions of TBT are designed to educate on, prepare for, and practice the four different types of exposure techniques. The next five sessions are focused on practicing and refining exposure practices as participants work through their lists of avoided situations/sensation/thoughts. The final session reviews treatment progress and relapse prevention strategies.

DSTs Control Condition Matching and Assignment To provide an evidence-based comparison for the TBT condition, DSTs will be used that are matched to the participant's most severe diagnosis, based upon the average of the ADIS interference and distress scores. If the scores are equivalent for two or more diagnoses, participants will be asked to list which diagnosis/symptoms that they find most impairing. DSTs will be included for each of the three targeted diagnoses, including PTSD (Cognitive Processing Therapy for PTSD), PD/AG (Cognitive Behavioral Therapy for PD/AG), and MDD (Cognitive Behavioral Therapy for MDD). Each of these DSTs have published manuals for administration and have received extensive support in the literature (Barlow, 2014). All three DSTs have been shown to improve comorbid symptomatology and therefore may be a more accurate comparison to TBT as compared to other available DSTs that may have less effect on comorbidity (e.g., applied relaxation for PD/AG).

Assessment of Psychiatric Symptomatology, and Treatment Satisfaction The battery of self-report questionnaires and a diagnostic interview will be completed pre-, mid-, and post-treatment and at the 6-month follow-up to track participants' progression through treatment and maintenance. To reduce the likelihood of missing data, all assessments will be scheduled separately from normal treatment sessions. Assessments of disorder-specific symptomatology, as well general symptoms of the depressive/anxiety disorders and related impairments, were chosen due to the transdiagnostic focus of the proposed study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be Veterans
* Participants must be clearly competent to provide informed consent for research participation
* Participants must meet DSM-5 criteria for panic disorder, major depressive disorder, or posttraumatic stress disorder
* Participants must be 18-80 years old

Exclusion Criteria:

* recent history (< 2 months) of psychiatric hospitalization or a suicide attempt as documented in their medical record or reported during clinical interview
* acute, severe illness or medical condition that likely will require hospitalization and/or otherwise interfere with study procedures as documented in their medical record (e.g., active chemotherapy/radiation treatment for cancer),
* recent start of new psychiatric medication (< 4 weeks)
* diagnosis of moderate-to-severe traumatic brain injury in their medical record and/or endorsement of screener questionnaire
* additional comorbid psychiatric diagnoses that were not listed as exclusion criteria are permitted as long as they are considered secondary to the principal diagnosis of MDD, PTSD, or PD/AG as determined by the diagnostic interview
* ineligible Veterans will be referred for non-study-related treatments within mental health at the RHJ VAMC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Gros, PhD MA BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon consultation with the local VA R&D and MUSC IRB committees after publication of primary research questions, the de-identified database will be made available to the public via the publishing journal's website (where applicable) as well as on (yet to be determined/selected) research community websites designed for the sharing of scientific findings and data.
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication of the primary outcome papers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transdiagnostic Behavior Therapy | Disorder Specific Therapies
Started | 153 | 151
Completed | 90 | 87
Not Completed | 63 | 64

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transdiagnostic Behavior Therapy | Disorder Specific Therapies | Total
Number analyzed (Participants) | 153 | 151 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.03 (14.34) | 42.57 (12.72) | 44.31 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 108 | 154
  Male | 107 | 43 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 53 | 62 | 115
  White | 89 | 82 | 171
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses DSM-5 criteria PTSD symptoms. Items are scored on a 5-point scale, range from 0 (not at all) to 4 (extremely). The total scale score ranges from 0 to 80 with higher scores associated with more severe symptomatology. Previous versions of the PCL have been shown to have excellent internal consistency and excellent test-retest reliability in Veterans. In addition, the PCL-5 has been incorporated into standard assessment for PTSD at the VA. The PCL5 will be used to assess symptoms of PTSD.
Time Frame: change from baseline to week 6 to week 12 to 6-month followup
Population: Numbers varied across time points due to missing data and participant discontinuation of psychotherapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdiagnostic Behavior Therapy | Disorder Specific Therapies
Number analyzed (Participants) | 136 | 129
score on a scale
  baseline | 48.0 (16.80) | 46.37 (16.12)
  mid-treatment: number analyzed (Participants) | 68 | 75
  mid-treatment | 42.44 (18.83) | 36.95 (19.18)
  post-treatment: number analyzed (Participants) | 61 | 65
  post-treatment | 35.00 (21.48) | 27.36 (19.04)
  follow-up: number analyzed (Participants) | 47 | 54
  follow-up | 37.40 (20.24) | 33.50 (20.00)

2. Primary Outcome: Patient Health Questionnaire - 9 (PHQ-9)
Description: The Patient Health Questionnaire - 9 (PHQ-9) is a 9-item depression scale derived from the Patient Health Questionnaire to assess the symptoms and diagnosis of depression. Items are scored on a 4-point scale, range from 0 (not at all) to 3 (nearly every day). The total scale score ranges from 0 to 27 with higher scores associated with more severe symptomatology. The PHQ-9 has been shown to have good reliability as well as validity in clinical samples. In addition, the PHQ-9 has been incorporated into standard screenings at the VA. The PHQ-9 will be used to assess symptoms of MDD.
Time Frame: change from baseline to week 6 to week 12 to 6-month followup
Population: Numbers varied across time points due to missing data and participant discontinuation of psychotherapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdiagnostic Behavior Therapy | Disorder Specific Therapies
Number analyzed (Participants) | 141 | 132
score on a scale
  baseline | 17.29 (5.66) | 16.28 (5.97)
  mid-treatment: number analyzed (Participants) | 72 | 75
  mid-treatment | 13.49 (6.70) | 12.87 (5.79)
  post-treatment: number analyzed (Participants) | 61 | 64
  post-treatment | 11.44 (6.82) | 10.32 (6.18)
  follow-up: number analyzed (Participants) | 45 | 49
  follow-up | 13.93 (7.31) | 13.84 (6.32)

3. Primary Outcome: Panic Disorder Severity Scale (PDSS)
Description: The Panic Disorder Severity Scale (PDSS) is a 7-item scale for the frequency and distress of panic attacks and related symptoms. Items are scored on a 5-point scale, range from 0 (no symptoms) to 4 (extreme symptoms). The total scale score ranges from 0 to 28 with higher scores associated with more severe symptomatology. The scale has demonstrated good internal consistency, test-retest reliability, and sensitivity to change during the course of treatment . The PDSS will be used to assess symptoms of PD/AG.
Time Frame: change from baseline to week 6 to week 12 to 6-month followup
Population: Numbers varied across time points due to missing data and participant discontinuation of psychotherapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transdiagnostic Behavior Therapy | Disorder Specific Therapies
Number analyzed (Participants) | 136 | 125
score on a scale
  baseline | 13.40 (6.48) | 12.59 (7.58)
  mid-treatment: number analyzed (Participants) | 68 | 74
  mid-treatment | 11.53 (7.03) | 11.25 (7.90)
  post-treatment: number analyzed (Participants) | 60 | 64
  post-treatment | 9.86 (7.98) | 6.98 (7.05)
  follow-up: number analyzed (Participants) | 51 | 59
  follow-up | 9.82 (7.98) | 8.81 (7.34)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 9 months
Arm/Group | Transdiagnostic Behavior Therapy | Disorder Specific Therapies
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/151
Serious Adverse Events (participants affected / at risk) | 1/153 | 2/151
Other Adverse Events (participants affected / at risk) | 13/153 | 8/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdiagnostic Behavior Therapy (N=153) | Disorder Specific Therapies (N=151)
psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 2 (2)
EMS call - Emergency Visit (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdiagnostic Behavior Therapy (N=153) | Disorder Specific Therapies (N=151)
Patient cancelled appt due to minor physical health complaints (e.g., stomach virus) (Psychiatric disorders) | 13 (20) | 8 (11)

LIMITATIONS AND CAVEATS:
Due to COVID-19 pandemic safety protocols, all procedures were completed via telehealth technologies with paper documentation exchanged via the United States Postal Service in accordance with VA pandemic-related research policies from November 2020 to September 2023, at which point procedures were transitioned to electronic delivery (e.g., REDCap) and in-person appointments (when requested) for the remainder of the study. These procedures resulted in higher than expected rates of missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT04293341/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT04293341/ICF_000.pdf